CLINICAL TRIAL: NCT03532347
Title: SharkCore Biopsy Needle Versus Standard FNA Needle in the Diagnosis of Solid Pancreatic Masses a Randomised Controlled Cross-over Trial of EUS Guided Tissue Acquisition - The SharkBITE Study
Brief Title: Endoscopic Ultrasound Guided Tissue Sampling (The SharkBITE Study)
Acronym: SharkBITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8090
Record Dates: First submitted 2017-11-01; First posted 2018-05-22 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm, Benign; Chronic Pancreatitis; Pancreas Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: All participants will receive both interventions the order i.e. FNB first or FNA first will be randomised. The pathologists reporting the samples will be blinded to the results with the alternative device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EUS tissue sampling (Experimental): Device: EUS-FNA needle (Beacon) 3 passes 25g needle from head of pancreas; 22g needle from neck, body and tail
  Device:EUS-FNB needle (Beacon Sharkcore) 3 passes 25g needle from head of pancreas; 22g needle from neck, body and tail
  Interventions: Device: EUS-FNA needle (Beacon)

INTERVENTIONS:
Device: EUS-FNA needle (Beacon) — Participants will be randomised to an initial 3 passes with Beacon FNA and then Beacon SharkCore biopsy needles or vice versa. 25g needles will be used for trans duodenal puncture and 22g for trans gastric puncture.
  Other Names: EUS-FNB needle (Beacon SharkCore)

SUMMARY:
This study compares the diagnostic performance of Endoscopic ultrasound (EUS) guided fine needle aspiration and EUS guided core biopsy (SharkCore) in patients with a solid pancreatic mass.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) guided fine needle aspiration (FNA) and fine needle biopsy (FNB) are the standard methods for obtaining tissue samples from tumours of the pancreas. The diagnostic accuracy by strict criteria is around 75-80%. A non diagnostic sample causes delay and the need for a repeat procedure. To date no significant difference has been found between standard FNA and standard FNB needles. A novel opposing bevel design (SharkCore) needle for FNB may provide better diagnostic performance. The aim of this study is to compare the performance of a standard needle and the Sharkcore needle. Patients attending for routine biopsy of a suspected pancreatic tumour will be invited to participate. All participants will have 3 samples taken with each needle. The samples from each needle will be processed and reported separately with the pathologists blinded as to the report from the other needle. Following the procedure participants will be observed as normal in the recovery area and allowed home later. Further study participation is limited to 1 telephone call at 7 days. Participants will be asked if they have developed any new symptoms since the procedure and whether they have had to seek medical attention for this.The risks of the study procedure are the same as those of a non study procedure. Both needle types are in routine use in our unit. The study will be performed in the endoscopy unit of the Freeman hospital. The study is funded by a grant from Medtronic the company who make the Sharkcore needle. The study is planned to recruit 108 participants over 10 months with a further 6 months of follow up. If the new needle is found to perform better its routine use will potentially reduce the delay experienced by patients as well as the cost incurred by repeat procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years and above with a solid pancreatic mass of any size, needing to Undergo the EUS examination to collect sample for diagnosis will be recruited for the study. The definition of a solid pancreatic mass will be based on an ultrasound or a CT scan result or based on the findings of a EUS examination done prior.
* Patients should have the ability and be willing to give informed consent

Exclusion Criteria:

* Cysts that do not have a significant solid component will be excluded
* Any contraindication to pancreatic biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
The sensitivity of standard Beacon FNA needle compared with the SharkCore (FNB) core biopsy needle in the sampling of solid pancreatic mass lesions. | During EUS procedure
  The sensitivity of standard Beacon FNA needle compared with the SharkCore (FNB) core biopsy needle in the sampling of solid pancreatic mass lesions during the EUS procedure.

SECONDARY OUTCOMES:
To compare the adequacy of the sample obtained with standard Beacon FNA needle compared with the SharkCore core biopsy needle in the sampling of solid pancreatic mass lesions. | During EUS Procedure
  To compare the adequacy of the sample obtained with standard Beacon FNA needle compared with the SharkCore core biopsy needle in the sampling of solid pancreatic mass lesions during EUS procedure per patient
Duration of pathologist reporting time | Per sample anticipated to be 1-2 weeks
  During pathologist diagnostic routine reporting period per sample standard is usually 1-2 weeks
Cost benefit analysis of the needle types | Over study period which is anticipated to be around 1 year
  An analysis to assess which needle is the most cost-effective
Duration of sampling procedures | During the EUS procedure
  Duration of sampling procedures during EUS procedure per patient

CONTACTS AND LOCATIONS:
Overall Officials: Kofi Oppong, Dr, Principal Investigator — Consultant Gastroenterologist
Locations (1):
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle, Newcastle Upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided